CLINICAL TRIAL: NCT01079884
Title: Gastroesophageal Reflux Disease, Sleep, and the Relationship to Driving Simulator Performance
Brief Title: Gastroesophageal Reflux Disease (GERD)/Nighttime Heartburn and Driving Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David A. Johnson, MD (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, David A. Johnson, MD, MD, Digestive & Liver Disease Specialists
Organization: Digestive & Liver Disease Specialists (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRUSESOM0438; 08-03-FB-0036 (Other: IRB)
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: esomeprazole 40 mg — 40 mg daily for 4 weeks
  Other Names: Nexium

SUMMARY:
The implications of sleep as it relates to the physiology and pathogenesis of a number of diseases has until recently been ignored. With the evolution of sleep laboratories, there is an emerging recognition of the relationship between sleep and various gastrointestinal diseases- in particular gastroesophageal reflux disease (GERD).( 1-5) It seems intuitive that waking/daytime activities or events may affect sleep and that any consequent sleep dysfunction may reciprocally further affect daytime function

DETAILED DESCRIPTION:
The implications of sleep as it relates to the physiology and pathogenesis of a number of diseases has until recently been ignored. With the evolution of sleep laboratories, there is an emerging recognition of the relationship between sleep and various gastrointestinal diseases in particular gastroesophageal reflux disease (GERD). Twenty five (25) patients meeting entry criteria will be compared with 25 matching historical control patients who do not have GERD symptoms or sleep disturbance. Patients will record heartburn symptoms and GERD-associated sleep disturbances on a diary card. These patients will be evaluated for baseline functionality GERD symptom scores, PSQI, driving simulator, bed partner questionnaire (optional) and receive 40 mg daily of Nexium® for 4 weeks. Primary outcome variable driving simulator performance will be the relief of nighttime heartburn during the last 7 days of the trial as recorded by the patient on a diary card. Secondary outcome variables include change from baseline to week 4 in the PSQI score, percentage of patients with complete resolution of sleep disturbances, relief of sleep disturbances, and percentage of days without GERD-associated sleep disturbances. Assessment of patients with complete resolution of daytime, night times, and 24-hour heartburn symptoms, and the percentage of patients with relief of daytime and 24-hour heartburn symptoms. The driving simulator performance will be compared at baseline and after 4 weeks of therapy with Nexium®. Also, where available, the bed partner PSQI will be compared at baseline and following treatment of the primary patient with Nexium® for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-60
* Diagnosis of GERD
* Nighttime heartburn

Exclusion Criteria:

* Less than 18 years old or older than 60 years of age
* Any conditions other than GERD that could be the primary cause of or a factor in your sleep disturbance. These include but are not limited to: severe anxiety, severe depression, panic attacks, sleep apnea, blocked airways, chronic pulmonary disease requiring oxygen therapy
* Restless leg syndrome
* Excessive need for nighttime urination (more than 2 times per night)
* Insomnia
* Excessive caffeine use (more than 4 standard 8-oz cups of coffee or caffeinated beverages, or 2 12-oz caffeinated sodas per day) or within 3 hours of sleep time
* Buerger's disease
* Use of a proton pump inhibitor
* Active gastrointestinal bleeding
* Severe, unresolved or unstable illnesses that the investigator feels would interfere with your participation in the study
* Severe liver disease
* Chronic illness that may cause excessive fatigue or low energy level such as chronic fatigue syndrome, or uncontrolled thyroid disease
* Need for anticoagulation therapy such as warfarin
* Active chemo or radiation therapy for cancer
* Prior gastric by-pass surgery
* History of seizures and/or anti-seizure medications (such as phenytoin or mephenytoin)
* Known hypersensitivity to esomeprazole or antacid tablets such as Tums, or Rolaids
* A history of drug addiction or alcohol abuse within the previous year
* Pregnant or lactating
* HIV+ status

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Driving impairment effects measured by the driving simulator (variance of 1.5 feet is abnormal). | 4 weeks
  All parameters will be assessed by both per protocol and intention to treat assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive and Liver Disease Specialists, Norfolk, Virginia, United States